CLINICAL TRIAL: NCT02971631
Title: The Effect of Glucagon Like Peptide-1 (GLP-1) on Glycaemic Profile and Eating Behaviour Following Gastrectomy
Brief Title: Gastrectomy, Eating Behaviour and GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Geoffrey Roberts, Clinical Research Associate, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A094265; 218762 (Other: IRAS)
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Gastric Cancer; Dumping Syndrome
Keywords: Dumping syndrome; Gastrectomy; GLP-1; Insulin
MeSH Terms: conditions — Stomach Neoplasms; Dumping Syndrome; Insulin Resistance | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Infusion of 1% human albumin in normal saline.
  Interventions: Other: Placebo
- Exendin (Experimental): Infusion of Exendin 9-39 in 1% human albumin in normal saline
  Interventions: Other: Exendin 9-39

INTERVENTIONS:
Other: Exendin 9-39 — Complete blockade of action of endogenous GLP-1 by Exendin 9-39. Defined as a physiological study, not a clinical trial as such (as advised by the UK MHRA).
  Arms: Exendin
Other: Placebo — Infusion of 1% human albumin in normal saline
  Arms: Placebo

SUMMARY:
Patients who have undergone gastrectomy (removal of the stomach) to treat or prevent cancer are known to have a significantly reduced quality of life. To date, there is very little information on the physiological causes of this. The investigators suspect that overproduction of a hormone (chemical) called glucagon like peptide-1 (GLP-1) released by the lining of the gut may play a role in the reduced appetite, weight loss and low blood sugar symptoms seen in this group. To investigate this, the investigators will study the response of 16 patients who have previously had a gastrectomy to a glucose drink, and a meal, while receiving an infusion of a specific blocker of GLP-1 or placebo. The investigators will examine the levels of sugar and associated hormones in the blood, food consumption and food reward behaviour using standard tools.

Participants will be invited to attend the Clinical Research Facility at Addenbrooke's Hospital for a screening visit, and two whole day study visits. The study has been designed to assess the role of overproduction of GLP-1 by completely blocking its actions, rather than assess the use of the blocking compound as a medication, and is therefore regarded as a physiological study, not a clinical trial.

The goal of this study is to demonstrate the magnitude of effect of GLP-1 on blood sugar and appetite derangement in patients who have had a gastrectomy. This will guide future work on the development of novel treatment paradigms for the post-gastrectomy patient group.

ELIGIBILITY:
Inclusion Criteria:

* • At least 3 months post completion of treatment for gastric cancer, or prophylactic gastrectomy

  * Aged at least 18 years
  * Able to tolerate an oral glucose tolerance test
  * Able to understand and retain all information regarding the study and give informed consent.
  * Willing to receive an infusion of human albumin solution

Exclusion Criteria:

* • Have a diagnosis of diabetes

  * Have a history of untreated anaemia in the last 3 months
  * Be aged under 18 years
  * Have active gastric cancer
  * Be pregnant or attempting to conceive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2018-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Roberts, MA BM BCh, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants recruited from Hereditary Diffuse Gastric Cancer patient population
Groups:
- Placebo Then Exendin: Infusion of 1% human albumin in normal saline on day one of study. Infusion of Exendin 9-39 in 1% human albumin in normal saline on day two of study (bolus of 7500pmol/kg followed by infusion of 500pmol/kg/minute for 4 hours).
- Exendin Then Placebo: Infusion of Exendin 9-39 in 1% human albumin in normal saline on day one of study (bolus of 7500pmol/kg followed by infusion of 500pmol/kg/minute for 4 hours).
  Infusion of 1% human albumin in normal saline on day two of study.
Period: First Intervention - One Day
Arm/Group | Placebo Then Exendin | Exendin Then Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Second Intervention - One Day
Arm/Group | Placebo Then Exendin | Exendin Then Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants were randomised to reveal both interventions, so baseline characteristics are reported for the whole study population.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Nadir Blood Glucose
Description: Lowest blood sugar reading during an oral glucose tolerance test while receiving infusion of GLP-1 antagonist. Please note participants will receive infusion of active compound for a maximum of four hours, with no expected effect of compound persisting for more than 30 minutes post-infusion.
Time Frame: As assessed during a 50g glucose tolerance test while receiving infusion of GLP-1 antagonist. At time 30-120 minutes of infusion of Exendin 9-39.
Population: Crossover study - analysis by paired T test
Measure: Mean (Standard Error); unit: mmol/l
Groups:
- Exendin: Infusion of Exendin 9-39 in 1% human albumin in normal saline
  Exendin 9-39: Complete blockade of action of endogenous GLP-1 by Exendin 9-39.
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
mmol/l | 3 (0.3) | 4.4 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Exendin; Test type: Superiority; p = 0.008, t-test, 2 sided; Paired analysis

2. Secondary Outcome: Total Insulin Secretion
Description: 60 minute incremental area under the curve (i.e. total) insulin secretion during 50g oral glucose tolerance test while receiving infusion of GLP-1 antagonist. Please note participants will receive infusion of active compound for a maximum of four hours, with no expected effect of compound persisting for more than 30 minutes post-infusion.
Time Frame: Samples collected at 0, 15, 30, 45 and 60 minutes post oral glucose tolerance test.
Measure: Mean (Standard Error); unit: pmol*minute/l
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
pmol*minute/l | 41000 (10400) | 14500 (2600)
Statistical Analysis 1: Comparison: Placebo vs Exendin; Test type: Superiority; p = 0.03, t-test, 2 sided; Paired analysis

3. Secondary Outcome: Eating Rate During ad Libitum Meal
Description: As measured by universal eating monitor, total weight of a standardised meal consumed over a measured time in grams per minute.
Time Frame: 150-210 minutes during infusion of Exendin 9-39 or placebo.
Measure: Mean (Standard Error); unit: grams/minute
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
grams/minute | 0.62 (0.12) | 0.66 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Exendin; For meal consumption rate; Test type: Superiority; p = 0.79, t-test, 2 sided; Paired analysis

4. Secondary Outcome: Decreased Hunger and Satiety Ratings During and After ad Libitum Meal
Description: Will be measured on visual analogue scale and reported as a score out of 100. Higher value indicated more hunger and more satiety.
Time Frame: 150-240 minutes during infusion of Exendin 9-39 or placebo and for 4 hours post-cessation of infusion.
Population: Unfortunately it proved impossible to collect data on hunger and fullness during the ad libitum meal, due to the cognitive effects of the gastrectomy which all of this group had undergone, meaning participants were unwilling to accurately record these sensations while eating. This data is therefore meaningless and was not analysed.
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Altered Food Attention.
Description: Food motivation can be measured by response rates to visual cues while being distracted by food related images. Will be measured with and without GLP-1 blockade to investigate effects of GLP-1 on food attention behaviour. Measure is of difference in response time when visual cue is colocated with a food related image vs a non-food related image, indicating degree of bias in attention to food images. Measure is undertaken during infusion at four timepoints - baseline (i.e. fasting), post oral glucose tolerance test (post-OGTT), before a standard meal (pre-meal) and after the meal (post-meal).
Time Frame: 0-240 minutes during infusion of Exendin 9-39 or placebo, assessed on four occasions (baseline or T0, post-OGTT, pre-meal, post-meal) using a validated dot-probe visual response tool and reported in response time (milliseconds).
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
milliseconds
  Time 0 | 17.9 (8.6) | 11.1 (7.1)
  Post OGTT | 18.2 (4.1) | 12.0 (9.0)
  Pre-meal | 24.8 (10.8) | 17.9 (8.9)
  Post-meal | 25.7 (10.8) | 10.7 (3.0)
Statistical Analysis 1: Comparison: Placebo vs Exendin; Baseline; Test type: Superiority; p = 0.20, t-test, 2 sided; Paired analysis
Statistical Analysis 2: Comparison: Placebo vs Exendin; Post-OGTT; Test type: Superiority; p = 0.58, t-test, 2 sided; Paired analysis
Statistical Analysis 3: Comparison: Placebo vs Exendin; Pre-meal; Test type: Superiority; p = 0.39, t-test, 2 sided; Paired analysis
Statistical Analysis 4: Comparison: Placebo vs Exendin; Post-meal; Test type: Superiority; p = 0.20, t-test, 2 sided; Paired analysis

6. Secondary Outcome: Altered Food Motivation
Description: Participant motivation to view particular food based cues is assessed by grip strength exerted to maintain those cues. Measure is undertaken during infusion at four timepoints - baseline (i.e. fasting), post oral glucose tolerance test (post-OGTT), before a standard meal (pre-meal) and after the meal (post-meal).
Time Frame: 0-240 minutes during infusion of Exendin 9-39 or placebo (baseline or T0, post-OGTT, pre-m, assessed on four occasions using a validated grip strength surrogate of food motivation and measured as the area under the curve of a grip force monitoring curve.
Measure: Mean (Standard Error); unit: Newton seconds
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
Newton seconds
  T0 / Baseline | 508 (182) | 219 (69)
  Post-OGTT | 139 (63) | 274 (56)
  Pre-meal | 328 (82) | 339 (116)
  Post-meal | 207 (82) | 227 (116)
Statistical Analysis 1: Comparison: Placebo vs Exendin; Baseline; Test type: Superiority; p = 0.26, t-test, 2 sided; Paired analysis
Statistical Analysis 2: Comparison: Placebo vs Exendin; Post-OGTT; Test type: Superiority; p = 0.06, t-test, 2 sided — Paired analysis
Statistical Analysis 3: Comparison: Placebo vs Exendin; Pre-meal; Test type: Superiority; p = 0.95, t-test, 2 sided; Paired analysis
Statistical Analysis 4: Comparison: Placebo vs Exendin; Post-meal; Test type: Superiority; p = 0.88, t-test, 2 sided; Paired analysis

7. Secondary Outcome: Number of Participants With Infusion Related Adverse Events as Assessed by CTCAE v4
Time Frame: 24 hours from onset of infusion.
Measure: Number; unit: participants
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Exendin; Test type: Superiority; p = 1, Other; 0 events over whole study, no statistical test appropriate

8. Secondary Outcome: Total Meal Consumption
Description: Total consumption amount of a standard meal during study intervention, measured in grams using a universal eating monitor.
Time Frame: 150-210 minutes during infusion of Exendin 9-39 or placebo
Measure: Mean (Standard Error); unit: grams
Arm/Group | Placebo | Exendin
Number analyzed (Participants) | 5 | 5
grams | 422 (45) | 434 (162)
Statistical Analysis 1: Comparison: Placebo vs Exendin; Test type: Superiority; p = 0.84, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 week.
Arm/Group | Placebo | Exendin
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT02971631/Prot_SAP_000.pdf